CLINICAL TRIAL: NCT00275678
Title: A Phase III Randomized, Multicenter Trial Comparing G-CSF Mobilized Peripheral Blood Stem Cell With Marrow Transplantation From HLA Compatible Unrelated Donors.
Brief Title: Comparison of Peripheral Blood Stem Cell Transplantation With Bone Marrow Transplantation for the Treatment of Serious Hematological Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other); University of Minnesota (Other); University of Florida (Other); Duke University (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Shakila Khan, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2158-03
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Blood Stem Cell Transplant

INTERVENTIONS:
Procedure: Blood stem cell versus bone marrow transplant — 1. Cyclophosphamide and Total Body Irradiation (CY-TBI)-based regimens that include at least 120 mg/kg cyclophosphamide and at least 1200 cGy of fractionated TBI.
  2. Busulfan and cyclophosphamide (BU-CY)-based regimens that include at least 14 mg/kg busulfan orally or 11.2 mg/kg busulfan intravenously (14 x 0.8 correction factor) or a targeted busulfan dosing strategy aimed at a serum concentration greater than 600 ng/mL at steady state and at least 120 mg/kg cyclophosphamide.
  3. Fludarabine and melphalan (Flu-Mel)-based regimens that include a fludarabine dose of least 120 mg per m2 and a melphalan dose of at least 140 mg per m2.
  4. Fludarabine, busulfan, and ATG (Flu-Bu-ATG)-based regimens that include a fludarabine dose of at least 120 mg/m2, at least 8 mg/kg busulfan orally or 250 mg/m2 busulfan intravenously, and at least 40 mg/kg equine ATG or 4 mg/kg rabbit ATG. Institutional standards should be followed for targeting plasma levels.

SUMMARY:
This study will compare the outcomes of study participants who have had peripheral blood stem cell transplantation or with those who have had bone marrow transplantation from an unrelated donor for the treatment of serious hematological malignancies.

DETAILED DESCRIPTION:
This study is a randomized, open-label, multicenter, prospective, comparative trial of granulocyte colony stimulating factor (G-CSF) mobilized peripheral blood stem cells verses marrow from unrelated donors for transplantation in patients with hematologic malignancies. The study will be comparing two-year survival probabilities between process has many steps after a matched donor is found. The donor also needs to give permission to join this study. Participants will be randomized to either peripheral blood stem cells (PBSC) or bone marrow. The kind of transplant the participant receives is random. Neither the participant nor the doctor may choose the type of transplant.

Participants will receive vaccinations for diphtheria, tetanus, hepatitis B and pneumococcus. Blood samples will be drawn as part of a participant's normal care. Blood samples will also be collected to see if infection fighting cells are working. These samples will be collected at 12 weeks, one year and then yearly until three years post transplant. Information will be collected from the participant's medical history. Participants will also have phone interviews conducted and questions will be asked about their physical and emotional health. Participants taking part in this study may be followed for up to 5 years.

ELIGIBILITY:
Participants may be eligible if they are between the ages of 18 to 66 years and are undergoing unrelated blood stem cell transplantation for the first time for the treatment of their hematological malignancy. Additional eligibility criteria will be gathered and evaluated by the transplant physician to determine if an individual is eligible to take part.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Two-year survival | 2 years
  The primary objective is to compare two-year survival probabilities between patients in the two study arms using an intent-to-treat analysis

SECONDARY OUTCOMES:
Two-year survival | 2 Years
  Transplanted patients randomized to the two study arms will be compared for the following endpoints: survival, incidences of neutrophil and platelet engraftment, graft failure, acute graft-versus-host disease (GVHD), chronic GVHD, time off all immunosuppressive therapy, relapse, infections, adverse events, immune reconstitution, and quality of life. Donors in each arm of the study will be compared for time to return to baseline toxicity score, CBC and WBC differential values after donation and quality of life.
Neutrophil Engraftment > 500/mcl | 2 Years
Primary graft failure | 2 years
Platelet engraftment > 20,000 and 50,000/mcl transfusion independent | 2 years
Acute GVHD of grades II-IV and III-IV | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Shakila P. Khan, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States